CLINICAL TRIAL: NCT02279485
Title: A Randomized, Open-Label, Crossover Study to Demonstrate Bioequivalence Between a 12-mg Dose of an Oral Suspension Formulation of Perampanel and a 12-mg Tablet Formulation of Perampanel Under Fasted and Fed Conditions in Healthy Subjects
Brief Title: A Study to Demonstrate Bioequivalence Between a 12-mg Dose of an Oral Suspension Formulation of Perampanel and a 12-mg Tablet Formulation of Perampanel Under Fasted and Fed Conditions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-A001-048
Record Dates: First submitted 2014-10-15; First posted 2014-10-31 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects; Bioequivalence; Fasted; Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perampanel - Group 1 (Experimental): Treatment A: Single oral dose of a 12-mg perampanel tablet under fasted condition.
  Treatment B: Single 12 mg dose of perampanel oral suspension under fasted condition.
  Subjects will be randomized on Study Day 1 for Treatment Period 1 to Treatment A or Treatment B. On Study Day 43 the subject will then receive the alternate Treatment for Treatment Period 2.
  Interventions: Drug: Perampanel
- Perampanel - Group 2 (Experimental): Treatment C: Single oral dose of a 12-mg perampanel tablet co-administered with high fat meal.
  Treatment D: Single 12 mg dose of perampanel oral suspension co-administered with high fat meal.
  Subjects will be randomized on Study Day 1 for Treatment Period 1 to Treatment C or Treatment D. On Study Day 43 the subject will then receive the alternate Treatment for Treatment Period 2.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel

SUMMARY:
This is an open-label, 2-arm, single-dose, randomized crossover study. The study will enroll a total of 100 subjects (2 arms with 50 subjects in each arm). In Arm 1, bioequivalence between the oral suspension and tablet formulations of perampanel will be evaluated under fasted conditions; in Arm 2, bioequivalence between the oral suspension and tablet formulations will be evaluated under fed conditions. In both study arms, subjects will be randomized on Study Day 1 for Treatment Period 1 to receive a single 12-mg dose for perampanel as either oral suspension or a tablet, and will then receive the alternative treatment on Study Day 43 of Treatment Period 2. Drug administration will be separated by a washout of at least 6 weeks between the two treatment periods.

ELIGIBILITY:
Inclusion Criteria

1. Healthy males or females, ages 18 to 55 years, inclusive, at the time of informed consent.
2. Body mass index (BMI) of 18 to 32 kg/m2, inclusive at Screening.
3. Females must not be lactating or pregnant at Screening or Baseline.
4. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, a doublebarrier method [such as condom plus diaphragm with spermicide], have a vasectomized partner with confirmed azoospermia, or an intrauterine device, contraceptive implant, or oral contraceptive that does not contain levogesterol) throughout the entire study period and for 30 days after study drug discontinuation. Females using hormonal contraceptives containing levogesterol must be on another form of contraception (such as double barrier method.) as well. If currently abstinent, the subject must agree to use a doublebarrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e. bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).

Exclusion Criteria

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical attention within 4 weeks of dosing.
2. Evidence of disease that may influence the outcome of the study within 4 weeks of dosing, eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system, or subjects who have a congenital abnormality in metabolism.
3. Any history of gastrointestinal surgery that may affect PK profiles of perampanel, eg, hepatectomy, nephrotomy, cholecystectomy, digestive organ resection or any gastrointestinal procedure for the purpose of weight loss (including Lapband), which would slow gastric emptying.
4. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening or Baseline.
5. Any laboratory abnormalities considered clinically significant by the investigator.
6. A prolonged QT/QTc interval (QTc greater than 450 msec) as demonstrated upon repeat ECG at Screening or Baseline.
7. History of prolonged QT/QTc interval.
8. History of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
9. History of ischemic heart disease (eg, acute coronary syndromes, stable angina), syncope or cardiac arrhythmias.
10. Siting heart rate less than 40 or greater than 100 beats/min at Screening or Baseline Period 1 and sitting systolic blood pressure greater than 140 mmHg or less than 90 mmHg or diastolic blood pressure greater than 90 mmHg or less than 60 mmHg at Screening or Baseline.
11. Hemoglobin less than 11.5 g/dLfor females and less than 12.5 g/dL for males at screen and Baseline check-in Period 1.
12. Subjects who experienced a weight loss or gain of greater than 10% between Screening and before dosing.
13. Subjects who received blood products within 4 weeks, donated blood within 8 weeks, or donated plasma within 1 week of dosing.
14. Hypersensitivity to the study drug or any of its excipients.
15. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening.
16. Known to be human immunodeficiency virus (HIV) positive at Screening.
17. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening.
18. History of use of illegal (or legalized) recreational drugs in the past year.
19. History of drug or alcohol dependency or abuse within approximately the last 2 years or who have a positive urine drug test or breath alcohol test at Screening or Baseline.
20. Engagement in strenuous exercise within 2 weeks before dosing (eg, marathon runners, weight lifters).
21. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days preceding informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Perampanel: AUC(0-t) | Up to 504 hours postdose in each treatment period
Pharmacokinetics of Perampanel: AUC(0-inf) | Up to 504 hours postdose in each treatment period
Pharmacokinetics of Perampanel: Cmax | Up to 504 hours postdose in each treatment period

SECONDARY OUTCOMES:
Pharmacokinetics of Perampanel: AUC(0-72h) | Up to 504 hours postdose in each treatment period
Pharmacokinetics of Perampanel: tmax | Up to 504 hours postdose in each treatment period
Pharmacokinetics of Perampanel: tlag | Up to 504 hours postdose in each treatment period
Pharmacokinetics of Perampanel: Lambda-z | Up to 504 hours postdose in each treatment period
Pharmacokinetics of Perampanel: t1/2 | Up to 504 hours postdose in each treatment period